CLINICAL TRIAL: NCT00543439
Title: An Open-label Study To Evaluate Prophylaxis Treatment, And To Characterize The Efficacy, Safety, And Pharmacokinetics Of B-domain Deleted Recombinant Factor Viii Albumin Free (Moroctocog Alfa [Af-cc]) In Children With Hemophilia A
Brief Title: Study Evaluating Prophylaxis Treatment & Characterizing Efficacy, Safety, & PK Of B-Domain Deleted Recombinant FVIII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3082B2-313; B1831001 (Other: Alias Study Number); 2006-005575-17 (EudraCT Number)
Record Dates: First submitted 2007-10-11; First posted 2007-10-15 (Estimated); Results first posted 2019-01-11 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2018-12

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — recombinant factor VIII SQ; F8 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): On-Demand therapy for 6 months, followed by Routine Prophylaxis treatment for 1 year.
  Interventions: Biological: Moroctocog alfa (AF-CC)
- 2 (Experimental): Routine Prophylaxis Crossover
  Interventions: Biological: Moroctocog alfa (AF-CC)

INTERVENTIONS:
Biological: Moroctocog alfa (AF-CC) — On-demand therapy for 6 months, followed by routine prophylaxis 25 IU/kg, administered every other day for 1 year.
  Other Names: Xyntha
  Arms: 1
Biological: Moroctocog alfa (AF-CC) — Routine prophylaxis crossover:
  45 IU/kg, administered 2 times a week for 1 year followed by 25 IU/kg administered every other day for 1 year, or, 25 IU/kg, administered every other day for 1 year, followed by 45 IU/kg, administered 2 times a week for 1 year.
  Other Names: Xyntha
  Arms: 2

SUMMARY:
The purpose of this research study is to determine the effectiveness, safety, and pharmacokinetics (PK) of moroctocog alfa (AF-CC) in previously treated subjects, who are younger than 6 years of age, with severe or moderately severe hemophilia A.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects, aged less than 6 years, with moderately severe to severe hemophilia A.
* A negative FVIII inhibitor titer at screening, and a medical history negative for a past FVIII inhibitor.
* At least 20 exposure days to any FVIII replacement product.
* Adequate hepatic and renal function
* CD4 count > 400 cells/uL, and if receiving antiviral therapy must be on a stable regimen

Additional criteria for subjects participating in the PK assessment:

* Male subjects as described immediately above except they must have a FVIII Activity of less than or equal to 1% confirmed by the central laboratory screening test
* Age < 6 years at time of PK assessment.
* The subject's size is sufficient to permit PK-related phlebotomy.
* The subject is able to comply with the procedures conducted during the PK assessment, including a mandatory 72-hour washout period preceding the PK assessment.

Exclusion Criteria:

* A history of FVIII inhibitor.
* Presence of a bleeding disorder in addition to hemophilia A.
* Treatment with any investigational drug or device within 30 days before the time of signing the informed consent form.
* Major or orthopedic surgery planned to occur during the course of the study.
* Regular (e.g., daily, every other day) use of antifibrinolytic agents or medications known to influence platelet function such as aspirin or certain nonsteroidal anti-inflammatory drugs (NSAIDs), or regular, concomitant therapy with immunomodulating drugs (e.g., intravenous immunoglobulin [IVIG], routine systemic corticosteroids).
* Known hypersensitivity to hamster protein.

Ages: 6 Months to 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 66 (Actual)
Dates: Start 2007-12 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (28):
- United States (7):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - OHSU Investigational Pharmacy, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Childrens Medical Center Dallas, Dallas, Texas
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Primary Children's Hospital, Salt Lake City, Utah
- Fundacion de la Hemofilia, Buenos Aires, Argentina
- Medizinische Universitaet Wien, Vienna, Austria
- Liga Colombiana de Hemofílicos y otras Deficiencias Sanguíneas, Bogotá, Colombia
- Clinical Hospital Centre Split, Split, Croatia
- Jordan University of Science and Technology, King Abdullah University Hospital, Irbid, Jordan
- Mexico (3):
  - Hospital Civil de Guadalajara Dr. Juan I. Menchaca, Guadalajara, Jalisco
  - Hospital y Clinica OCA S.A. de C.V., Colonia Centro, Monterrey, Nuevo LEON
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
- New Zealand (2):
  - Christchurch Hospital, Christchurch, South Island
  - Canterbury District Health Board, Christchurch
- Sultan Qaboos University Hospital, Muscat, Oman
- Centro Medico Monte Carmelo, Urbanización La Victoria, Arequipa, Peru
- Samodzielny Publiczny Dzieciecy Szpital Kliniczny, Warsaw, Poland
- Sanador, Bucharest, Romania
- Turkey (Türkiye) (7):
  - Cukurova University Tip Fakultesi, Balcali/Adana, Adana
  - Ege Universitesi Tip Fakultesi Cocuk Hastanesi, Izmir, Bornova
  - Istanbul Universtesi Istanbul Tip Fakultesi, Çapa, Istanbul
  - On Dokuz Mayis University Faculty of Medicine, Samsun, Kurupelit
  - Akdeniz Universitesi Tip Fakultesi, Antalya
  - Dr. Behcet Uz Child and Diseases And Surgery Education and Research Hospital, Izmir
  - Erciyes Universitesi Tip Fakultesi, Kayseri

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3082B2-313&StudyName=Study%20Evaluating%20Prophylaxis%20Treatment%20%26%20Characterizing%20Efficacy%2C%20Safety%2C%20%26%20PK%20Of%20B-Domain%20Deleted%20Recombinant%20FVIII

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants for 1 of the sites, were excluded from efficacy and safety analysis due to data integrity issues, however were reported in participant flow and baseline analysis.
Groups:
- Moroctocog Alfa (AF-CC),OD Cohort:OD Therapy Then RP Therapy: Participants who consented for pharmacokinetic assessment received single 50 international units per kilogram [IU/kg] infusion of AF-CC on Day 1 prior start of study treatment.Period 1:participants were treated with on-demand (OD) therapy intravenous (IV) infusion of AF-CC for 6 months(Day 1 up to Month 6)prescribed by investigator based on current recommendations for OD therapy with licensed product Xyntha (Minor bleeding:repetition of IV infusion of AF-CC,20-40 IU/kg,every 12-24 hours (hr) until resolved for at least 1 day,depending upon severity of bleeding episode;Moderate bleeding:repetition of IV infusion of AF-CC,30-60 IU/kg,every 12-24 hr for 3-4 days/until adequate local hemostasis achieved;Major bleeding:repetition of IV infusion of AF-CC,60-100 IU/kg,every 8-24 hr until bleeding resolved).Then in Period 2 participants received IV infusion of AF-CC at 25 IU/kg once in 2 days up to 12 months (Month 7 to Month 18) as RP therapy and if required were treated with OD IV infusion.
- Moroctocog Alfa(AF-CC),RP Cohort:RP 25 IU/kg Then RP 45IU/kg: Participants received a single 50 IU/kg infusion of moroctocog alfa (AF-CC) on Day 1 before initiation of moroctocog alfa (AF-CC) study treatment either in on demand cohort or routine prophylaxis cohort. In Period 1 participants for routine prophylaxis therapy, received IV infusion of moroctocog alfa (AF-CC) at 25 IU/kg once in 2 days up to 12 months (Day 1 up to Month 12). Period 1 was followed by Period 2 where participants received IV infusion of moroctocog alfa (AF-CC) at 45 IU/kg, twice per week up to 12 months (Month 13 up to Month 24) as routine prophylaxis therapy. Participants were treated OD IV infusion up to 12 months.
- Moroctocog Alfa(AF-CC), RP Cohort:RP 45 IU/kg Then RP25IU/kg: Participants received a single 50 IU/kg infusion of moroctocog alfa (AF-CC) on Day 1 before initiation of moroctocog alfa (AF-CC) study treatment either in on demand cohort or routine prophylaxis cohort. In Period 1 participants for routine prophylaxis therapy, received IV infusion of moroctocog alfa (AF-CC) at 45 IU/kg twice per week up to 12 months (Day 1 up to Month 12). Period 1 was followed by Period 2 where participants received IV infusion of moroctocog alfa (AF-CC) at 25 IU/kg, once in 2 days up to 12 months (Month 13 up to Month 24) as routine prophylaxis therapy. Participants were treated OD IV infusion up to 12 months.
Period: Period 1
Arm/Group | Moroctocog Alfa (AF-CC),OD Cohort:OD Therapy Then RP Therapy | Moroctocog Alfa(AF-CC),RP Cohort:RP 25 IU/kg Then RP 45IU/kg | Moroctocog Alfa(AF-CC), RP Cohort:RP 45 IU/kg Then RP25IU/kg
Started | 10 | 29 | 27
Treated | 9 | 29 | 27
Completed | 9 | 26 | 25
Not Completed | 1 | 3 | 2
Not completed — Adverse Event | 0 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1
Period: Period 2
Arm/Group | Moroctocog Alfa (AF-CC),OD Cohort:OD Therapy Then RP Therapy | Moroctocog Alfa(AF-CC),RP Cohort:RP 25 IU/kg Then RP 45IU/kg | Moroctocog Alfa(AF-CC), RP Cohort:RP 45 IU/kg Then RP25IU/kg
Started | 9 | 26 | 25
Completed | 8 | 25 | 23
Not Completed | 1 | 1 | 2
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (mITT) analysis population included all participants for whom a legal acceptable representative had signed the informed consent/assent form and who received at least 1 dose of moroctocog alfa (AF-CC).
Groups:
- Total: Total of all reporting groups
Arm/Group | Moroctocog Alfa (AF-CC),OD Cohort:OD Therapy Then RP Therapy | Moroctocog Alfa(AF-CC),RP Cohort:RP 25 IU/kg Then RP 45IU/kg | Moroctocog Alfa(AF-CC), RP Cohort:RP 45 IU/kg Then RP25IU/kg | Total
Number analyzed (Participants) | 9 | 29 | 27 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.7 (1.05) | 4.4 (1.84) | 4.1 (2.28) | 4.3 (1.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 9 | 29 | 27 | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 8 | 24 | 22 | 54
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 5 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Mean Annualized Bleed Rate (ABR) by Treatment: On Demand Cohort
Description: ABR for each participant was calculated as the number of bleeds requiring administration of moroctocog alfa (AF-CC) divided by the total therapy duration (in days), then multiplied by 365.25 (days in a year).
Time Frame: Day 1 up to Month 6 (OD Cohort, OD Therapy, Period 1); Month 7 up to Month 18 (OD Cohort, RP 25 IU/kg, Period 2)
Population: Intent-to-treat (ITT) analysis population included all participants for whom a legal acceptable representative had signed the informed consent/assent form. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Bleeds per year
Groups:
- Moroctocog Alfa (AF-CC), On Demand Cohort: On Demand Therapy: In Period 1, participants for on-demand therapy were treated with IV infusion of moroctocog alfa (AF-CC) for 6 months (Day 1 up to Month 6) as prescribed by the investigator based on current recommendations for on-demand treatment with licensed product Xyntha (Minor bleeding: repetition of IV infusion of Moroctocog alfa, 20-40 IU/kg, every 12-24 hours as necessary until resolved for at least 1 day, depending upon severity of bleeding episode; Moderate bleeding: repetition of IV infusion of Moroctocog alfa, 30-60 IU/kg, every 12-24 hours for 3-4 days or until adequate local hemostasis was achieved; Major bleeding: repetition of IV infusion of moroctocog alfa (AF-CC), 60-100 IU/kg, every 8-24 hours until bleeding was resolved).
- Moroctocog Alfa (AF-CC), On Demand Cohort: RP Therapy 25 IU/kg: In Period 2, participants for on-demand cohort received IV infusion of moroctocog alfa (AF-CC) at 25 IU/kg once in 2 days up to 12 months (Month 7 up to Month 18) as routine prophylaxis therapy.
Arm/Group | Moroctocog Alfa (AF-CC), On Demand Cohort: On Demand Therapy | Moroctocog Alfa (AF-CC), On Demand Cohort: RP Therapy 25 IU/kg
Number analyzed (Participants) | 9 | 8
Bleeds per year | 47.0 (32.2) | 1.5 (2.2)
Statistical Analysis 1: Comparison: Moroctocog Alfa (AF-CC), On Demand Cohort: On Demand Therapy vs Moroctocog Alfa (AF-CC), On Demand Cohort: RP Therapy 25 IU/kg; Ratio of the arithmetic means of the ABR for OD cohort: OD therapy to OD cohort: RP therapy 25 IU/kg was calculated. One-sided 95% CI for this ratio was reported; Test type: Superiority; p = 0.0020, Paired t-test; Ratio of arithmetic means = 0.03, 95% CI 1-sided [upper limit 0.08]

2. Secondary Outcome: Mean Annualized Bleed Rate (ABR) by Treatment: Routine Prophylaxis Cohort
Description: as for outcome 1
Time Frame: Day 1 up to Month 24 (RP Cohort, Period 1 and Period 2)
Population: ITT analysis population included all participants for whom a legal acceptable representative had signed the informed consent/assent form. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Bleeds per year
Groups:
- Moroctocog Alfa (AF-CC), RP Cohort: RP Therapy 45 IU/kg: Participants of routine prophylaxis cohort, received IV infusion of moroctocog alfa (AF-CC) at 45 IU/kg, twice per week up to 12 months as routine prophylaxis therapy each for either Period 1 (Day 1 up to Month 12) or Period 2 (Month 13 up to Month 24) of the study.
- Moroctocog Alfa (AF-CC), RP Cohort: RP Therapy 25 IU/kg: Participants of routine prophylaxis cohort, received IV infusion of moroctocog alfa (AF-CC) at 25 IU/kg, once in 2 days up to 12 months as routine prophylaxis therapy for either Period 1 (Day 1 up to Month 12) or Period 2 (Month 13 up to Month 24) of the study.
Arm/Group | Moroctocog Alfa (AF-CC), RP Cohort: RP Therapy 45 IU/kg | Moroctocog Alfa (AF-CC), RP Cohort: RP Therapy 25 IU/kg
Number analyzed (Participants) | 38 | 38
Bleeds per year | 3.3 (5.3) | 2.2 (4.1)
Statistical Analysis 1: Comparison: Moroctocog Alfa (AF-CC), RP Cohort: RP Therapy 45 IU/kg vs Moroctocog Alfa (AF-CC), RP Cohort: RP Therapy 25 IU/kg; Test type: Equivalence — 90% 2-sided CI for the mean difference in ABRs for the 2 prophylaxis regimens for ITT participants was constructed using the t distribution with n-1 degrees of freedom (n equals the number of participants) to assess the equivalence of the 2 regimens. Equivalence was demonstrated and the null hypothesis rejected if the limits of the 90% CI fell wholly within the interval of (-4, 4) bleeds per year; Mean Difference (Final Values) = 1.1, 90% CI 2-sided [0.03 to 2.22]

3. Secondary Outcome: Mean of Moroctocog Alfa (AF-CC) Infusions Administered To Treat Bleeding Episode: All Participants
Description: In this outcome measure, the mean of total number of moroctocog alfa (AF-CC) on-demand infusions administered to treat each bleeding episode was reported, regardless of participant cohort or period during which it occurred.
Time Frame: Day 1 up to Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Infusions
Units Other Than Participants: bleed
Groups:
- Moroctocog Alfa (AF-CC): All Participants: All participants who received moroctocog alfa-(AF-CC) 50 IU/kg for PK assessment on Day 1 prior start of study treatment and as on demand or routine prophylaxis treatment (25 and 45 IU/kg).
Arm/Group | Moroctocog Alfa (AF-CC): All Participants
Number analyzed (Participants) | 38
Number analyzed (bleed) | 562
Infusions | 1.5 (1.38)

4. Secondary Outcome: Number of Treated Bleeds Classified on Basis of Response to First Infusion of Moroctocog Alfa (AF-CC) as On-Demand Treatment: OD Therapy (OD and RP Cohort)
Description: Number (no.) of bleeds treated are reported on basis of response to first infusion of study drug, at 4-point scale: excellent, good, moderate, no response. Excellent:definite pain relief and/or improvement in bleeding signs within 8 hours (hr) after infusion, no additional infusion administered; Good:definite pain relief and/or improvement in bleeding signs within 8 hr after infusion, at least 1 additional infusion administered for complete resolution or with no additional infusion administered; Moderate:probable or slight improvement starting after 8 hr following infusion,at least 1 additional infusion administered for complete resolution; No Response: no improvement at all between infusions or during 24 hr interval following infusion or condition worsen. Bleeds for which response not recorded, reported as:Data Not Recorded. Total no. of first infusions may not be equal to total no. of bleeds if bleed was: missing start date/dose information or treated initially with non-study FVIII.
Time Frame: Day 1 up to Month 24
Population: as for outcome 2
Measure: Number; unit: Bleeds
Units Other Than Participants: bleeds
Groups:
- Moroctocog Alfa (AF-CC): On Demand Therapy: Participants of either on demand cohort or routine prophylaxis cohort were treated for bleeds, as needed on demand, with IV infusion of moroctocog alfa (AF-CC) up to 24 months as prescribed by the investigator based on current recommendations for on-demand treatment with licensed product Xyntha (Minor bleeding: repetition of IV infusion of moroctocog alfa (AF-CC), 20-40 IU/kg, every 12-24 hours as necessary until resolved for at least 1 day, depending upon severity of bleeding episode; Moderate bleeding: repetition of IV infusion of moroctocog alfa (AF-CC), 30-60 IU/kg, every 12-24 hours for 3-4 days or until adequate local hemostasis was achieved; Major bleeding: repetition of IV infusion of moroctocog alfa (AF-CC), 60-100 IU/kg, every 8-24 hours until bleeding was resolved).
Arm/Group | Moroctocog Alfa (AF-CC): On Demand Therapy
Number analyzed (Participants) | 38
Number analyzed (bleeds) | 559
Bleeds
  Excellent | 376
  Good | 150
  Moderate | 27
  No Response | 2
  Data Not Recorded | 4

5. Secondary Outcome: Number of Treated Spontaneous Bleeds by Time Interval Between Bleed Onset and Prior Moroctocog Alfa (AF-CC) Prophylaxis Dose: Routine Prophylaxis Therapy
Description: In this outcome measure number of treated spontaneous bleeds are reported according to the time interval between bleed onset and prior moroctocog alfa (AF-CC) routine prophylaxis dose. Following time intervals used to report this outcome measure: lesser than or equal to (<=) 24 hours, greater than (>) 24 hours to <=48 hours, >48 hours to <=72 hours, >72 hours. For reporting arm: "Moroctocog alfa (AF-CC),OD and RP Cohort: RP Therapy 25 IU/kg" cumulative data for routine prophylaxis cohort (Day 1 up to Month 24, Period 1 and Period 2) and on demand cohort (Month 7 up to Month 18, Period 2) is reported.
Time Frame: Day 1 up to Month 24 (RP Cohort, RP 25 IU/kg and 45 IU/kg, Period 1 and 2); Month 7 up to Month 18 (OD Cohort, RP 25 IU/kg, Period 2)
Population: Analysis population included all participants for whom a legal acceptable representative had signed the informed consent/assent form and who reported a spontaneous bleeding episode following a routine prophylaxis dose.
Measure: Number; unit: Bleeds
Units Other Than Participants: bleeds
Groups:
- Moroctocog Alfa(AF-CC),OD and RP Cohort: RP Therapy 25 IU/kg: Participants of routine prophylaxis cohort received IV infusion of moroctocog alfa (AF-CC) at 25 IU/kg, once in 2 days up to 12 months as routine prophylaxis therapy each for either Period 1 (Day 1 up to Month 12) or Period 2 (Month 13 up to Month 24) of the study. And participants of on demand cohort for Period 2 of the study, received IV infusion of moroctocog alfa (AF-CC) at 25 IU/kg, once in 2 days as routine prophylaxis therapy up to 12 months (Month 7 up to Month 18).
Arm/Group | Moroctocog Alfa (AF-CC), RP Cohort: RP Therapy 45 IU/kg | Moroctocog Alfa(AF-CC),OD and RP Cohort: RP Therapy 25 IU/kg
Number analyzed (Participants) | 9 | 7
Number analyzed (bleeds) | 28 | 18
Bleeds
  <=24 hours | 1 | 3
  >24 hours to <=48 hours | 4 | 6
  >48 hours to <=72 hours | 10 | 2
  >72 hours | 13 | 7

6. Secondary Outcome: Number of Participants Requiring Prophylaxis Regimen Escalation: Routine Prophylaxis Therapy
Description: During prophylaxis, criteria for prophylaxis regimen escalation are the occurrence, over a 4-week duration (and in the absence of a confirmed FVIII inhibitor), of (a) 2 or more spontaneous bleeds into a major joint and/or target joint, or (b) 3 or more spontaneous bleeds (consisting of joint bleeds and/or significant soft tissue/muscle or other site bleeds). If either criterion was met, the participant was escalated to a more intense prophylaxis regimen of 45 IU/kg, administered every other day. Participant who meet dose escalation criteria while on prophylaxis regimen of 45 IU/kg, were escalated to a higher intensity regimen designated by the investigator. Significant spontaneous bleeds were those that led to a transient or persistent loss of function. For reporting arm: "Moroctocog alfa (AF-CC),OD and RP Cohort: RP Therapy 25 IU/kg", cumulative data for RP cohort (Day 1 up to Month 24, Period 1 and Period 2) and OD cohort (Month 7 up to Month 18, Period 2) is reported.
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Moroctocog Alfa (AF-CC), RP Cohort: RP Therapy 45 IU/kg | Moroctocog Alfa(AF-CC),OD and RP Cohort: RP Therapy 25 IU/kg
Number analyzed (Participants) | 39 | 48
Participants | 2 | 1

7. Secondary Outcome: Mean Routine Prophylaxis Dose (IU/kg) of Moroctocog Alfa (AF-CC) Received: Routine Prophylaxis Therapy
Description: Mean RP dose (by weight) for each participant was calculated as his total moroctocog alfa (AF-CC) consumption (in IU) divided by weight (in kg). For reporting arm: "Moroctocog alfa (AF-CC),OD and RP Cohort: RP Therapy 25 IU/kg", cumulative data for routine prophylaxis cohort (Day 1 up to Month 24, Period 1 and Period 2) and on demand cohort (Month 7 up to Month 18, Period 2) is reported.
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: IU/kg
Groups:
- Moroctocog Alfa(AF-CC), On Demand Cohort: RP Therapy 25IU/kg: In Period 2, participants of on demand cohort, received IV infusion of moroctocog alfa (AF-CC) at 25 IU/kg once in 2 days up to 12 months (Month 7 up to Month 18) as routine prophylaxis therapy.
Arm/Group | Moroctocog Alfa(AF-CC), On Demand Cohort: RP Therapy 25IU/kg | Moroctocog Alfa (AF-CC), RP Cohort: RP Therapy 45 IU/kg | Moroctocog Alfa (AF-CC), RP Cohort: RP Therapy 25 IU/kg | Moroctocog Alfa(AF-CC),OD and RP Cohort: RP Therapy 25 IU/kg
Number analyzed (Participants) | 8 | 39 | 40 | 48
IU/kg | 25 (4.6) | 46 (5.8) | 26 (5.4) | 26 (5.2)

8. Secondary Outcome: Mean of Total Number Moroctocog Alfa (AF-CC) Infusions Received: Routine Prophylaxis Therapy
Description: In this outcome measure mean of total number of infusions of moroctocog alfa (AF-CC) received by participant is reported. For reporting arm: "Moroctocog alfa (AF-CC),OD and RP Cohort: RP Therapy 25 IU/kg", cumulative data for routine prophylaxis cohort (Day 1 up to Month 24, Period 1 and Period 2) and on demand cohort (Month 7 up to Month 18, Period 2) is reported.
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Infusions
Arm/Group | Moroctocog Alfa(AF-CC), On Demand Cohort: RP Therapy 25IU/kg | Moroctocog Alfa (AF-CC), RP Cohort: RP Therapy 45 IU/kg | Moroctocog Alfa (AF-CC), RP Cohort: RP Therapy 25 IU/kg | Moroctocog Alfa(AF-CC),OD and RP Cohort: RP Therapy 25 IU/kg
Number analyzed (Participants) | 8 | 39 | 40 | 48
Infusions | 170 (31.3) | 91 (22.4) | 150 (37.0) | 154 (36.6)

9. Secondary Outcome: Mean of Total Number of Days Participants Exposed to Moroctocog Alfa (AF-CC): Routine Prophylaxis Therapy
Description: For reporting arm: "Moroctocog alfa (AF-CC),OD and RP Cohort: RP Therapy 25 IU/kg", cumulative data for routine prophylaxis cohort (Day 1 up to Month 24, Period 1 and Period 2) and on demand cohort (Month 7 up to Month 18, Period 2) is reported.
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Moroctocog Alfa(AF-CC), On Demand Cohort: RP Therapy 25IU/kg | Moroctocog Alfa (AF-CC), RP Cohort: RP Therapy 45 IU/kg | Moroctocog Alfa (AF-CC), RP Cohort: RP Therapy 25 IU/kg | Moroctocog Alfa(AF-CC),OD and RP Cohort: RP Therapy 25 IU/kg
Number analyzed (Participants) | 8 | 39 | 40 | 48
Days | 170 (31.3) | 91 (22.3) | 150 (37.0) | 153 (36.5)

10. Secondary Outcome: Mean of Total Number of Infusions of Moroctocog Alfa (AF-CC) Received Per Week to Assess Compliance: Routine Prophylaxis Therapy
Description: Participants' compliance to their assigned prophylaxis regimen was measured by following: a) number of infusions received per week and b) dose received. In this outcome measure mean of total number of infusions of moroctocog alfa (AF-CC) received by participants per week is reported. For reporting arm: "Moroctocog alfa (AF-CC),OD and RP Cohort: RP Therapy 25 IU/kg" cumulative data for routine prophylaxis cohort (Day 1 up to Month 24, Period 1 and Period 2) and on demand cohort (Month 7 up to Month 18, Period 2) is reported.
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Infusions per week
Arm/Group | Moroctocog Alfa (AF-CC), RP Cohort: RP Therapy 45 IU/kg | Moroctocog Alfa(AF-CC),OD and RP Cohort: RP Therapy 25 IU/kg
Number analyzed (Participants) | 39 | 48
Infusions per week | 2.1 (0.81) | 3.3 (0.18)

11. Secondary Outcome: Terminal Phase Half Life (t1/2) of Factor VIII (FVIII) Activity
Description: Plasma decay half-life is the time measured for the FVIII activity to decrease by one half.
Time Frame: 0.5, 8, 24, 28 and 32 hours post dose on Day 1
Population: Analysis population included all participants for whom a legal acceptable representative had signed the informed consent/assent form, were in a non bleeding state, participated in a single pharmacokinetic (PK) assessment at the start of the study and for whom an adequate PK profile had been obtained.
Measure: Mean (Standard Deviation); unit: Hour
Groups:
- Moroctocog Alfa (AF-CC): 50 IU/kg: Participants received a single 50 IU/kg infusion of moroctocog alfa (AF-CC) on Day 1 before initiation of moroctocog alfa (AF-CC) study treatment either in on demand cohort or routine prophylaxis cohort.
Arm/Group | Moroctocog Alfa (AF-CC): 50 IU/kg
Number analyzed (Participants) | 7
Hour | 8.86 (2.3513)

12. Secondary Outcome: Clearance (CL) of Factor VIII Activity
Description: Clearance is a measure of the volume of plasma from which FVIII activity is removed per unit time. It was reported in units milliliter per hour per kilogram (mL/hr/kg).
Time Frame: 0.5, 8, 24, 28 and 32 hours post dose on Day 1
Population: Analysis population included all participants for whom a legal acceptable representative had signed the informed consent/assent form, were in a non bleeding state, participated in a single PK assessment at the start of the study and for whom an adequate PK profile had been obtained.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr/kg
Arm/Group | Moroctocog Alfa (AF-CC): 50 IU/kg
Number analyzed (Participants) | 7
mL/hr/kg | 5.822 (59)

13. Secondary Outcome: Incremental Recovery of Factor VIII Activity
Description: Incremental recovery was the increase in circulating FVIII activity for every international unit (IU) of moroctocog alfa (AF-CC) administered per kilogram of body weight of participant. It was measured in international units per deciliter per international units per kilogram ([IU/dL]/[IU/kg]).
Time Frame: Day 1, Month 6
Population: Analysis population included all participants for whom legal acceptable representative had signed informed consent/assent form, were in non-bleeding state, participated in single PK assessment at start of study and for whom an adequate PK profile had been obtained. "Number analyzed" signifies participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: (IU/dL)/(IU/kg)
Arm/Group | Moroctocog Alfa (AF-CC): 50 IU/kg
Number analyzed (Participants) | 7
(IU/dL)/(IU/kg)
  Day 1: number analyzed (Participants) | 6
  Day 1 | 1.4438 (0.6145)
  Month 6: number analyzed (Participants) | 2
  Month 6 | 1.4148 (0.4046)

14. Secondary Outcome: Maximum Concentration of Factor VIII Activity
Description: Maximum concentration of FVIII activity was measured in international units per milliliter (IU/mL).
Time Frame: 0.5, 8, 24, 28 and 32 hours post dose on Day 1
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/mL
Arm/Group | Moroctocog Alfa (AF-CC): 50 IU/kg
Number analyzed (Participants) | 7
IU/mL | 0.7005 (60)

15. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of Factor VIII Activity
Description: Area under FVIII activity-time profile from time zero extrapolated to infinite time. AUCinf is reported in units: international units*hour per milliliter (IU*hour/mL).
Time Frame: 0.5, 8, 24, 28 and 32 hours post dose on Day 1
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU*hr/mL
Arm/Group | Moroctocog Alfa (AF-CC): 50 IU/kg
Number analyzed (Participants) | 7
IU*hr/mL | 9.02 (50)

16. Secondary Outcome: Area Under the Curve From Time Zero to Last Measurable Concentration (AUClast) of Factor VIII Activity
Description: Area under the FVIII activity -versus-time curve from time zero to the time of the last quantifiable concentration.
Time Frame: 0.5, 8, 24, 28 and 32 hours post dose on Day 1
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU*hr/mL
Arm/Group | Moroctocog Alfa (AF-CC): 50 IU/kg
Number analyzed (Participants) | 7
IU*hr/mL | 8.04 (46)

17. Secondary Outcome: Steady-State Volume of Distribution (Vss) of Factor VIII Activity
Description: Volume of distribution is defined as the theoretical volume in which the total amount of FVIII would need to be uniformly distributed to produce the observed plasma concentration of FVIII. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state.
Time Frame: 0.5, 8, 24, 28 and 32 hours post dose on Day 1
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliter per kilogram
Arm/Group | Moroctocog Alfa (AF-CC): 50 IU/kg
Number analyzed (Participants) | 7
Milliliter per kilogram | 78.38 (50)

18. Secondary Outcome: Mean Residence Time (MRT) of Factor VIII Activity
Description: MRT was calculated as AUMCinf /AUCinf-TI/2, where AUMCinf is the area under the moment curve from time zero to infinity and TI is the duration of infusion.
Time Frame: 0.5, 8, 24, 28 and 32 hours post dose on Day 1
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Moroctocog Alfa (AF-CC): 50 IU/kg
Number analyzed (Participants) | 7
Hour | 13.46 (33)

19. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) According to Severity
Description: AE is untoward medical occurrence in clinical investigation participant administered product or medical device;event need not necessarily had causal relationship with treatment or usage.Treatment-emergent are events between first dose of study drug and up to 28 days after last dose of study drug (up to 25 months)that were absent before treatment or that worsened relative to pretreatment state.AEs were classified into following on basis of severity:1)mild = did not interfere with participant's usual function;2)moderate=interfered to some extent with participant's usual function;3)severe=interfered significantly with participant's usual function;4)life threatening=AE required discontinuation of study drug,participant was at immediate risk of death.All participants in study received AF-CC.AEs were not collected separately for each intervention for participants.All participants were properly combined for analysis,regardless of regimen were following at time,regardless of OD or RP cohort.
Time Frame: Day 1 up to Month 25
Population: Analysis population included all participants for whom a legal acceptable representative had signed the informed consent/assent form and were analyzed for safety. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Moroctocog Alfa (AF-CC): All Participants
Number analyzed (Participants) | 49
Participants
  Mild | 12
  Moderate | 29
  Severe | 8
  Life threatening | 0

20. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events
Description: A treatment related AE is any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event had a causal relationship with the treatment or usage. All participants in the study received moroctocog alfa-(AF-CC). Adverse events were not collected separately for each intervention for the participants. All participants were properly combined for the analysis and was regardless of the regimen they were following at the time, and regardless of OD or RP cohort.
Time Frame: Day 1 up to Month 25
Population: Analysis population included all participants for whom a legal acceptable representative had signed the informed consent/assent form and were analyzed for safety.
Measure: Count of Participants; unit: Participants
Arm/Group | Moroctocog Alfa (AF-CC): All Participants
Number analyzed (Participants) | 51
Participants | 49

21. Secondary Outcome: Number of Participants With Confirmed FVIII Inhibitor Development
Description: Confirmed FVIII inhibitors were defined as a neutralizing antibody to FVIII with a titer value of greater than or equal to (>=) 0.6 Bethesda units (BU) per millimeter in a sample assayed using the Nijmegen assay at the central laboratory.
Time Frame: Day 1 up to Month 24
Population: Analysis population included all participants for whom legal acceptable representative had signed informed consent/assent form and who received 1 dose of moroctocog alfa (AF-CC) and were at risk for confirmed FVIII inhibitor development.
Measure: Count of Participants; unit: Participants
Arm/Group | Moroctocog Alfa (AF-CC): All Participants
Number analyzed (Participants) | 49
Participants | 3

22. Secondary Outcome: Number of Participants With Incidence of Less Than Expected Therapeutic Effect (LETE): On Demand Therapy
Description: LETE occurs in OD setting if participant recorded 2 successive "No Response" (no improvement at all between infusions, or condition worsens) ratings after 2 successive infusions of study drug. Infusions must have been given within 24 hours (hr) of each other for treatment of same bleeding event in absence of confounding factors (known presence or subsequent identification of a FVIII inhibitor, known inadequate dose for type and/or severity of bleed in opinion of investigator, delay of >4 hr between onset of bleed to infusion, delay of >24 hr before administration of a follow-up infusion, known compromised study drug, faulty administration of study drug, participant had an underlying, predisposing condition responsible for bleed in opinion of investigator. For reporting arm: "Moroctocog alfa (AF-CC), OD and RP Cohort: RP Therapy 25 IU/kg", cumulative data for RP cohort (Day 1 up to Month 24, Period 1 and Period 2) and OD cohort (Month 7 up to Month 18, Period 2) is reported.
Time Frame: Day 1 up to Month 24 (RP Cohort, RP 25 IU/kg and 45 IU/kg, Period 1 and 2); Day 1 up to Month 6 (OD Cohort, OD Therapy, Period 1); Month 7 up to Month 18 (OD Cohort, RP 25 IU/kg, Period 2)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Moroctocog Alfa (AF-CC) OD Cohort: OD Therapy: In Period 1, participants of OD cohort, as OD therapy were treated with IV infusion of moroctocog alfa (AF-CC) for 6 months (Day 1 up to Month 6) as prescribed by the investigator based on current recommendations for on-demand treatment with licensed product Xyntha (Minor bleeding: repetition of IV infusion of AF-CC, 20-40 IU/kg, every 12-24 hours as necessary until resolved for at least 1 day, depending upon severity of bleeding episode; Moderate bleeding: repetition of IV infusion of AF-CC, 30-60 IU/kg, every 12-24 hours for 3-4 days or until adequate local hemostasis was achieved; Major bleeding: repetition of IV infusion of AF-CC, 60-100 IU/kg, every 8-24 hours until bleeding was resolved).
Arm/Group | Moroctocog Alfa (AF-CC) OD Cohort: OD Therapy | Moroctocog Alfa (AF-CC), RP Cohort: RP Therapy 45 IU/kg | Moroctocog Alfa(AF-CC),OD and RP Cohort: RP Therapy 25 IU/kg
Number analyzed (Participants) | 9 | 42 | 51
Participants | 0 | 0 | 0

23. Secondary Outcome: Number of Participants With Incidence of Less Than Expected Therapeutic Effect (LETE): Routine Prophylaxis Therapy
Description: LETE in prophylaxis setting if there was a spontaneous bleed within 48 hours after a regularly scheduled prophylactic dose of study drug (which was not used to treat a bleed) in the absence of confounding factors (known presence or subsequent identification of a FVIII inhibitor, known inadequate prophylactic dose [a dose less than that prescribed in participant's regimen], known lack of adherence to the prescribed prophylaxis regimen, bleed occurs in a target joint identified at the start of the study, known compromised study drug, faulty administration of study drug, participant had an underlying, predisposing condition responsible for the bleed in the opinion of the investigator. Therefore, LETE in the prophylaxis setting was the occurrence of a bleed. For reporting arm: "Moroctocog alfa (AF-CC), OD and RP Cohort: RP Therapy 25 IU/kg", cumulative data for RP cohort (Day 1 up to Month 24, Period 1 and Period 2) and OD cohort (Month 7 up to Month 18, Period 2) is reported.
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Moroctocog Alfa (AF-CC), RP Cohort: RP Therapy 45 IU/kg | Moroctocog Alfa(AF-CC),OD and RP Cohort: RP Therapy 25 IU/kg
Number analyzed (Participants) | 42 | 51
Participants | 3 | 5

ADVERSE EVENTS:
Time Frame: Day 1 up to Month 25
Description: Same event may appear both an AE and SAE.However,what is presented are distinct events.An event may be categorized as serious in 1 participant and as non-serious in another,or participant may have experienced both SAE and NSAE.All participants in study received moroctocog alfa(AF-CC).AEs were not collected separately for each intervention for participants.All participants were properly combined for analysis and was regardless of regimen they were following at time,regardless of OD or RP cohort.
Arm/Group | Moroctocog Alfa (AF-CC): All Participants
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 13/51
Other Adverse Events (participants affected / at risk) | 49/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Moroctocog Alfa (AF-CC): All Participants (N=51)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 2
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Torticollis (Musculoskeletal and connective tissue disorders) | 1
Factor VIII inhibition (Blood and lymphatic system disorders) | 3
Device related infection (Infections and infestations) | 2
Limb injury (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Monoplegia (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Haematoma (Vascular disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Catheter site rash (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Moroctocog Alfa (AF-CC): All Participants (N=51)
Upper respiratory tract infection (Infections and infestations) | 16
Nasopharyngitis (Infections and infestations) | 14
Influenza (Infections and infestations) | 8
Tonsillitis (Infections and infestations) | 7
Pharyngitis (Infections and infestations) | 5
Varicella (Infections and infestations) | 4
Viral infection (Infections and infestations) | 3
Pyrexia (General disorders) | 24
Fatigue (General disorders) | 4
Joint injury (Injury, poisoning and procedural complications) | 10
Limb injury (Injury, poisoning and procedural complications) | 10
Head injury (Injury, poisoning and procedural complications) | 7
Contusion (Injury, poisoning and procedural complications) | 5
Fall (Injury, poisoning and procedural complications) | 5
Face injury (Injury, poisoning and procedural complications) | 3
Laceration (Injury, poisoning and procedural complications) | 3
Traumatic haematoma (Injury, poisoning and procedural complications) | 3
Vomiting (Gastrointestinal disorders) | 10
Diarrhoea (Gastrointestinal disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 6
Toothache (Gastrointestinal disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 5
Tooth loss (Gastrointestinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10
Back pain (Musculoskeletal and connective tissue disorders) | 4
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 4
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 3
Headache (Nervous system disorders) | 7
Tooth extraction (Surgical and medical procedures) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2015-10-02): https://cdn.clinicaltrials.gov/large-docs/39/NCT00543439/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-30): https://cdn.clinicaltrials.gov/large-docs/39/NCT00543439/SAP_001.pdf